CLINICAL TRIAL: NCT00937924
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial of Promethazine and Diphenhydramine as Adjunct Sedatives for Endoscopic Ultrasound (EUS) and Endoscopic Retrograde Cholangiopancreatography (ERCP)
Brief Title: Adjunct Sedatives in Endoscopic Ultrasound (EUS) and Endoscopic Retrograde Cholangiopancreatography (ERCP) Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kenneth J. Chang, Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20075810
Record Dates: First submitted 2008-06-04; First posted 2009-07-13 (Estimated); Results first posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Endoscopic Ultrasound (EUS); Endoscopic Retrograde Cholangiopancreatography (ERCP)
Keywords: EUS; ERCP; Sedation Level; Adverse Symptoms; Recovery time
MeSH Terms: interventions — Meperidine; Midazolam; Diphenhydramine; Promethazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Meperidine and midazolam group (Placebo Comparator): Control. Normal Saline Injections.
  Interventions: Drug: Meperidine, Midazolam
- Meperidine and midazolam, plus Diphenhydramine group (Experimental): Diphenhydramine injections given as adjunct sedative.
  Interventions: Drug: Meperidine, Midazolam; Drug: Diphenhydramine
- Meperidine and midazolam, plus Promethazne group (Experimental): Promethazine given as an adjunct sedative.
  Interventions: Drug: Meperidine, Midazolam; Drug: Promethazine

INTERVENTIONS:
Drug: Meperidine, Midazolam
Drug: Diphenhydramine
  Arms: Meperidine and midazolam, plus Diphenhydramine group
Drug: Promethazine
  Arms: Meperidine and midazolam, plus Promethazne group

SUMMARY:
The purpose of this study is to compare meperidine/midazolam with diphenhydramine, meperidine/midazolam with promethazine, and meperidine/midazolam with placebo as sedation methods. The investigators are interested to see whether adjunct sedatives (diphenhydramine and promethazine) will improve sedation.

DETAILED DESCRIPTION:
Comparing sedation techniques during invasive endoscopic procedures such as ERCP and EUS is a relatively unexplored area of clinical research. In particular, the effectiveness of adjunct sedatives such as diphenhydramine and promethazine during ERCP/EUS procedures has not been studied. Achieving a moderate sedation level may be ideal for ERCP/EUS procedures in order to provide adequate patient comfort, amnesia, and completion of intended endoscopic procedures. The relevance of further studies in this area is apparent. In terms of clinical practice; over-sedation can lead to decreased airway protection, longer post-procedural recovery times, and unnecessary drug cost; under-sedation can lead to patient anxiety, agitation, recall, and longer procedural time.

ELIGIBILITY:
Inclusion Criteria:

* Willing participants between 18 and 75 years of age who present for ERCP or EUS at H.H. Comprehensive Chao Digestive Disease Center.

Exclusion Criteria:

* History of allergic or adverse reactions to midazolam, diphenhydramine, or promethazine.
* Acute asthma, narrow angle glaucoma, concurrent use of potent inhibitors of CYP3A4 (amprenavir, atazanavir, or ritonavir), pregnancy, or the inability to consent.
* Patients with conditions that preclude safe conscious sedation will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chang, MD, Principal Investigator — UC Irvine
Locations (1):
- H.H. Chao Comprehensive Digestive Disease Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Normal Saline: Control. Normal Saline Injections.
- 2 Diphenhydramine: Diphenhydramine injections given as adjunct sedative.
- 3 Promethzine: Promethazine given as an adjunct sedative.
Period: Overall Study
Arm/Group | 1 Normal Saline | 2 Diphenhydramine | 3 Promethzine
Started | 102 | 101 | 101
Completed | 58 | 57 | 60
Not Completed | 44 | 44 | 41
Not completed — Lost to Follow-up | 44 | 44 | 41

BASELINE CHARACTERISTICS:
Population: We had complete data available on 175 patients. The other patients had incomplete or missing data.
Groups:
- 1- Saline Control Group: Control. These patients will receive Normal Saline Injections to serve as controls.
  Saline: Saline solution injections
- 2 - Diphenhydramine Sedation Group: These patients will receive Diphenhydramine injections given as adjunct sedative.
  Diphenhydramine: Diphenhydramine injections
- 3 - Promethazine Sedation Group: Promethazine given as an adjunct sedative.
  Promethazine: Promethazine
- Total: Total of all reporting groups
Arm/Group | 1- Saline Control Group | 2 - Diphenhydramine Sedation Group | 3 - Promethazine Sedation Group | Total
Number analyzed (Participants) | 57 | 58 | 60 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 27 | 28 | 30 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (3) | 56 (3) | 58 (3) | 57 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 26 | 78
  Male | 31 | 32 | 34 | 97

OUTCOME MEASURES:

1. Primary Outcome: Average Percentage of Sedation Failures
Description: The percentage of participants who could not complete the procedure due inability to achieve proper sedation level
Time Frame: From onset of sedation to completion of procedure, approximately 1 hour.
Measure: Mean (Standard Deviation); unit: percentage of participants
Groups:
- 1 - Control Arm: Normal Saline Injections.: Control Arm: Normal Saline Injections.
  After placement of IV catheter and obtaining baseline vitals, including blood pressure, pulse, and oxygen saturation, subjects received pre-procedure injection of normal saline prior to standard sedation agents. The standard agents included standard doses of meperidine and midazolam, both administered via IV catheter and titrated under standard endoscopy protocol.
- 2 - Diphenhydramine Injections Given as Adjunct Sedative.: Diphenhydramine injections given as adjunct sedative.
  After placement of IV catheter and obtaining baseline vitals, including blood pressure, pulse, and oxygen saturation, subjects received pre-procedure injection of diphenhydramine prior to standard sedation agents. The standard agents included standard doses of meperidine and midazolam, both administered via IV catheter and titrated under standard endoscopy protocol.
- 3 - Promethazine Given as an Adjunct Sedative.: Promethazine given as an adjunct sedative.
  After placement of IV catheter and obtaining baseline vitals, including blood pressure, pulse, and oxygen saturation, subjects received pre-procedure injection of promethizine prior to standard sedation agents. The standard agents included standard doses of meperidine and midazolam, both administered via IV catheter and titrated under standard endoscopy protocol.
Arm/Group | 1 - Control Arm: Normal Saline Injections. | 2 - Diphenhydramine Injections Given as Adjunct Sedative. | 3 - Promethazine Given as an Adjunct Sedative.
Number analyzed (Participants) | 58 | 57 | 60
percentage of participants | 14 (2) | 13 (2) | 5 (1)

2. Primary Outcome: Time to Achieve Adequate Level of Sedation to Begin Procedure
Time Frame: Pre-Endoscopic Procedure (up to 1 hour maximum)
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- 1 - Control. Normal Saline Injections.: Control. Normal Saline Injections.
  Saline: Saline solution injections
- 2 - Diphenhydramine Injections Given as Adjunct Sedative.: Diphenhydramine injections given as adjunct sedative.
  Diphenhydramine: Diphenhydramine injections
- 3 - Promethazine Given as an Adjunct Sedative.: Promethazine given as an adjunct sedative.
  Promethazine: Promethazine
Arm/Group | 1 - Control. Normal Saline Injections. | 2 - Diphenhydramine Injections Given as Adjunct Sedative. | 3 - Promethazine Given as an Adjunct Sedative.
Number analyzed (Participants) | 58 | 57 | 60
minutes | 15 (3) | 13 (4) | 14 (5)

3. Primary Outcome: Time for Recovery
Time Frame: Post-Endoscopic Procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1 - Control. Normal Saline Injections. | 2 - Diphenhydramine Injections Given as Adjunct Sedative. | 3 - Promethazine Given as an Adjunct Sedative.
Number analyzed (Participants) | 58 | 57 | 60
minutes | 21.3 (5) | 29.5 (4) | 51.5 (6)

4. Secondary Outcome: Adverse Symptoms From Sedative Agents
Time Frame: Approximately 3 hours.
Measure: Mean (Standard Deviation); unit: adverse events
Arm/Group | 1 - Control. Normal Saline Injections. | 2 - Diphenhydramine Injections Given as Adjunct Sedative. | 3 - Promethazine Given as an Adjunct Sedative.
Number analyzed (Participants) | 58 | 57 | 60
adverse events | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Arm/Group | 1 - Control. Normal Saline Injections. | 2 - Diphenhydramine Injections Given as Adjunct Sedative. | 3 - Promethazine Given as an Adjunct Sedative.
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/57 | 0/60
Other Adverse Events (participants affected / at risk) | 0/58 | 0/57 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No